CLINICAL TRIAL: NCT03702218
Title: An Open-label Pilot Study to Determine the Safety and Efficacy of Hepatitis C Uninfected Recipients of Renal and Liver Transplants From a Currently Infected or Previously Infected Hepatitis C Donor
Brief Title: Hepatitis C Positive Donor Into Hepatitis C Negative Recipients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: never started
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00083009
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C
Keywords: Transplantation; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Hep C Ab + NAT - Donor to Naïve Recipient (Experimental): HCV Ab and HCV NAT testing at 3 days, week 1, week 2 and monthly for 3 months, at 6 months and 1 year. In approximately 16% of the patients, active hepatis C infection will ensue. For these patients, treatment is as follows.
  Liver Transplant:
  • Combinations of choice:
  * Mavyret (glecaprevir/pibrentasvir) - Genotype 1-6
  * Harvoni (ledipasvir/sofosbuvir) + Ribavirin - Genotypes 1, 4, 5, 6; GFR>30
  * Epclusa (sofosbuvir/velpatasvir) + Ribavirin - Genotypes 1-6; GFR>30
  Kidney Transplant:
  • Combinations of choice:
  * Mavyret (glecaprevir/pibrentasvir) - genotype 1-6
  * Harvoni (sofosbuvir/ledipasvir) - genotype 1, 4; GFR>30
  Interventions: Drug: Direct Acting Antivirals
- Hep C Ab+ NAT+ Donor to Naïve Recipient (Experimental): HCV RNA levels, liver biochemistries, and renal function will be measured 3 days after transplant. HCV Genotype will be determined after HCV RNA is >1,000 IU/mL. HCV RNA levels will be measured weekly after transplant until HCV treatment is initiated.
  Liver Transplant:
  • Combinations of choice:
  * Mavyret (glecaprevir/pibrentasvir) - Genotype 1-6
  * Harvoni (ledipasvir/sofosbuvir) + Ribavirin - Genotypes 1, 4, 5, 6; GFR>30
  * Epclusa (sofosbuvir/velpatasvir) + Ribavirin - Genotypes 1-6; GFR>30
  Kidney Transplant:
  • Combinations of choice:
  * Mavyret (glecaprevir/pibrentasvir) - genotype 1-6
  * Harvoni (sofosbuvir/ledipasvir) - genotype 1, 4; GFR>30
  Interventions: Drug: Direct Acting Antivirals
- Hep C Ab- NAT - Donor to Naïve Recipient (Active Comparator): Current standard of care for donor recipient infectious disease matching. No treatment necessary
  Interventions: Drug: Direct Acting Antivirals

INTERVENTIONS:
Drug: Direct Acting Antivirals — Patients who are given organ transplants from donors that are Ab positive and NAT negative or Ab positive and NAT positive for Hepatitis C will be treated with direct acting antivirals after transplant if they become NAT+ for hepatitis C.
  Interventions as follows.
  Liver Transplant:
  • Combinations of choice:
  * Mavyret (glecaprevir/pibrentasvir) - Genotype 1-6
  * Harvoni (ledipasvir/sofosbuvir) + Ribavirin - Genotypes 1, 4, 5, 6; GFR>30
  * Epclusa (sofosbuvir/velpatasvir) + Ribavirin - Genotypes 1-6; GFR>30
  Kidney Transplant:
  • Combinations of choice:
  * Mavyret (glecaprevir/pibrentasvir) - genotype 1-6
  * Harvoni (sofosbuvir/ledipasvir) - genotype 1, 4; GFR>30

SUMMARY:
Despite many efforts to increase the size of the donor pool, there is a large and growing disparity between the number of donor kidneys and livers available for transplantation and the number of patients on the transplant waiting list. New donor pools are needed to satisfy the lack of available donor organs, along with expanded criteria for the existing donor pools.

A new standard of care now exists at most local and regional transplant centers. This new standard of care is based on the use of multiple direct-acting antiviral agents (DAAs) for treatment of hepatitis C virus (HCV) that have been approved by the Food and Drug Administration (FDA) for the treatment of hepatitis C and are associated with high HCV cure rates and minimal side effect profiles. The efficacy and tolerability of these medications has allowed the expansion of the available donor pool by making HCV antibody positive non viremic organs and HCV-viremic organs (when HCV is detectable in the blood) available to HCV-naive recipients on the organ transplantation waiting list. Expansion of this donor pool may decrease time on the waiting list and improve quality of life and survival while waiting for organ transplantation.

Study Aim:

We propose a clinical protocol to utilize solid organs from exposed and/or HCV-viremic organ donors for transplantation into HCV negative recipients.

The primary purpose of the clinical protocol is to:

Collect prospective standard of care laboratory data on the results of these interventions

DETAILED DESCRIPTION:
Once the donor is accepted for transplantation and the recipient enrolled in the innovative clinical practice, donor HCV Ab status will be requested to initiate HCV RNA viral load testing.

Donor data will be recorded as per our standard practice and as mandated by UNOS. Our University of Maryland Medical Center team will be responsible for the donor operation as per standard of care.

Hep C Ab + NAT - Donor to Naïve Recipient This group will be monitored as illustrated in figure 1. Hep C Ab+ NAT+ Donor to Naïve Recipient HCV RNA levels, liver biochemistries, and renal function will be measured 3 days after transplant. HCV Genotype will be determined after HCV RNA is >1,000 IU/mL. HCV RNA levels will be measured weekly after transplant until HCV treatment is initiated.

Due to risk of HBV reactivation with DAA therapy, Hepatitis B surface antigen, surface antibody and core antibody status will be determined prior to HCV therapy. In patients with a prior exposure to HBV (i.e. positive HBV core antibody), Hepatitis B surface antigen levels will be monitored throughout therapy.

All patients will be seen in the Hepatology clinic within 4 weeks of transplant to establish care and follow-up.

HCV Therapy DAA therapy will be prescribed to all patients according to AASLD and IDSA joint guidelines, after giving consideration to the transplanted organ, renal function, and HCV genotype. All regimens exclude administration of ribavirin.

Therapy will be initiated as soon as possible (pending initiation of oral intake and insurance approval) following organ transplantation.

DAAs will be prescribed, after which medications will then be delivered to the patient's home or to the bedside.

If therapy is delayed beyond the 4-week appointment with Hepatology post-transplant, a protocol to monitor for infection, new-onset diabetes mellitus, glomerulonephritis and severe cholestatic hepatitis will be implemented. This protocol will include weekly blood work to include: CBC with differential, hepatic function panel, basic metabolic panel, and coagulation studies.

Liver Transplant:

• Combinations of choice:

* Mavyret (glecaprevir/pibrentasvir) - Genotype 1-6
* Harvoni (ledipasvir/sofosbuvir) + Ribavirin - Genotypes 1, 4, 5, 6; GFR>30
* Epclusa (sofosbuvir/velpatasvir) + Ribavirin - Genotypes 1-6; GFR>30

Kidney Transplant:

• Combinations of choice:

* Mavyret (glecaprevir/pibrentasvir) - genotype 1-6
* Harvoni (sofosbuvir/ledipasvir) - genotype 1, 4; GFR>30 HCV Follow-Up HCV RNA, complete blood count (CBC) and liver biochemistries will be checked 4 weeks, 8 weeks, and 12 weeks after starting therapy. In patients previously exposed to HBV, HBV surface antigen will be followed qualitatively at the same intervals.

HCV RNA will also be checked 12 weeks after completion of therapy to define cure, or sustained virologic response. As part of long-term follow-up, HCV RNA will be checked annually at routine post-transplant visits.

If SVR is not achieved, a second, and if needed, third antiviral regimen will be provided to the participant at no cost.

Transplant, Post-Operative, Immunosuppression Follow Up All will be as per UMMC standard of care. Unless otherwise contraindicated, tacrolimus immune suppression will be favored, due to drug-drug interactions associated with DATs and cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* RECIPIENT INCLUSION CRITERIA

  * Patients undergoing solid organ transplantation, including liver, kidney, and simultaneous liver-kidney who are not chronically infected with HCV
  * No evident contraindication for organ transplantation
  * HCV RNA negative (can be isolated HCV antibody positive provided the patient will have no history of previously treated HCV)
  * Age 18-75 years at the time of transplantation
  * Signed Informed Consent Form
  * No identified living organ donor
  * Able to travel to the University of Maryland for routine post-transplant and HCV follow-up visits
  * Men and women must agree to use at least one barrier method to prevent any secretion exchange
  * No active illicit drug use

DONOR INCLUSION CRITERIA

• Qualitative HCV nucleic acid test (NAT) positive and/or Hepatitis C antibody positive HCV donors offered to the University of Maryland.

Exclusion Criteria:

RECIPIENT EXCLUSION CRITERIA

* History of prior solid organ transplantation
* HIV infection
* HBV surface antigen or DNA positive. Organs from HCV positive donors who are also Hepatitis B core antibody positive (hepatitis B surface antigen negative) can be used. These patients will however need to undergo prophylaxis for HBV according to their respective organ specific criteria and during treatment for hepatitis C due to the increased risk of reactivation of hepatitis B with DAA therapy
* Waitlisted for a multi-organ transplant (with the exception of simultaneous liver-kidney transplant)
* HCV RNA positive (can be isolated HCV antibody positive provided the patient will have no history of previously treated HCV)
* Prior direct-acting antiviral (DAA) treatment for HCV. Patients previously treated with interferon-based regimens may be included.

DONOR EXCLUSION CRITERIA

* Every donor that is considered unsuitable by the transplant surgeon for any reason.
* Hepatocellular carcinoma
* HIV infection
* Use of HCV positive livers to be determined according to current existing criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
SVR after receiving an organ from a donor previously exposed to Hepatitis C after treatment direct-acting antiviral drugs. | 12 months
  To improve access to transplantation with use of HCV-non viremic and HCV-viremic organs in HCV negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in peer reviewed journals.
Supporting Information: SAP

REFERENCES:
- [Background] Goldberg DS, Blumberg E, McCauley M, Abt P, Levine M. Improving Organ Utilization to Help Overcome the Tragedies of the Opioid Epidemic. Am J Transplant. 2016 Oct;16(10):2836-2841. doi: 10.1111/ajt.13971. Epub 2016 Aug 24. PMID 27438538
- [Background] Bari K, Luckett K, Kaiser T, Diwan T, Cuffy M, Schoech MR, Safdar K, Blackard JT, Apewokin S, Paterno F, Sherman KE, Zucker SD, Anwar N, Shah SA. Hepatitis C transmission from seropositive, nonviremic donors to non-hepatitis C liver transplant recipients. Hepatology. 2018 May;67(5):1673-1682. doi: 10.1002/hep.29704. Epub 2018 Mar 26. PMID 29205441